CLINICAL TRIAL: NCT03888313
Title: Pretreatment Group Consultation for Patients With Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Eva Haglind, MD, PhD, professor, Principal Investigator Clinical Professor Eva Haglind, Sahlgrenska University Hospital
Other Study IDs: INFOM
Record Dates: First submitted 2019-03-16; First posted 2019-03-25 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-01

CONDITIONS: Colorectal Neoplasm
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients participating in the pretreatment group consultation: Patients who chosse to participate in a group consultation (with other patients also in the process of undergoing surgery for colorectal cancer).
  Interventions: Other: Pretreatment group consultation

INTERVENTIONS:
Other: Pretreatment group consultation — A consultation in group with several patients and one surgeon

SUMMARY:
An explorative study of the patients' experience of participating at a group consultation, together with other patients with newly diagnosed colon or rectal cancer

DETAILED DESCRIPTION:
The group consultation is planned to be on the Friday of the same week as the patient recieved a suggested treatment plan i.e. after MDT, at a personal consultation with his/her colorectal surgeon. During the group consultation the steps necessary for the patient to take responsability for in connection with the operation. Ample time for questions, clarifications and discussions. Appropriate clinical trials are presented

ELIGIBILITY:
Inclusion Criteria:

* Patients participating in the pretreatment group consultation

Exclusion Criteria:

* Not able to answer questionnaire

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colon or rectal cancer at the Sahlgrenska University Hospital/Östra planned for surgical treatment
Sampling Method: Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
The patient's experience of participating in a pretreatment group consultation | Before start of treatment
  A questionnaire with questions on the patient's experience of the information received and their experience of participating in the pretreatment group consultation will be used to collect descriptive data. Some of the questions have been developed through semi-structured interviews with patients with colon or rectal cancer other are standardized questionnaires used in other studies.
  The questionnaire includes questions on which information resources the patients have used (such as social media, patient organizations).Their experience of the pretreatment group consultation will be assessed by "Would you recommend someone in the same situation as you to attend the pretreatment group consultation?". Possible answering options are "Yes", "No" and "Don't know". The EuroQol's EQ-5D-5L for assessment of health related quality of will be included mainly as a tool for assurance of external validity, and not as an outcome measure. Both the indices and the VAS-scale may be used.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Angenete, MD, PhD, Study Chair — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital/Östra, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Walming S, Angenete E, Bock D, Block M, de la Croix H, Wedin A, Haglind E. Preoperative Group Consultation Prior to Surgery for Colorectal Cancer-an Explorative Study of a New Patient Education Method. J Cancer Educ. 2022 Oct;37(5):1304-1311. doi: 10.1007/s13187-020-01951-7. Epub 2021 Jan 14. PMID 33447870